CLINICAL TRIAL: NCT07106905
Title: Relationships Between Handgrip Strength, Physical Workload, Depression, and Low Back Pain in Mothers of Children With Disabilities Following COVID-19 Pandemic
Brief Title: Low Back Pain in Mothers of Children With Disabilities
Status: Completed | Type: Observational
Sponsor: Selvin BALKİ (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Sponsor-Investigator, Selvin BALKİ, Associate Professor, Ph.D., Cumhuriyet University
Organization: Cumhuriyet University (Other)
Other Study IDs: SCU-FTR-SBF-02
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Low back pain; Mothers of children with disabilities.; Handgrip strength; Physical workload; Depression
MeSH Terms: conditions — Low Back Pain; Depression | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mothers of children with disabilities
  Interventions: Other: Measurements

INTERVENTIONS:
Other: Measurements — These measurements are used in other clinical applications. However, the effectiveness of these measurements in discriminating the presence of low back pain in mothers of children with disabilities over the past year has been identified.

SUMMARY:
This is a cross-sectional study that aims to determine the prevalence of low back pain in mothers of children with disabilities following the COVID-19 pandemic and to describe its relationship with exposure to the virus, handgrip strength, physical workload, and depression.

DETAILED DESCRIPTION:
Low back pain is a very common problem in mothers of children with disabilities. Musculoskeletal pain have been on the rise with COVID-19 but the effects of the pandemic on the prevalence of low back pain in mothers of children with disabilities have not been investigated. The relationship between handgrip strength and low back pain is well known. There are limited studies investigating handgrip strength or muscle strength in mothers of children with disabilities, and no studies examining the relationship between handgrip strength and low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having a disabled child
* Being responsible for the care of a disabled child
* Having provided care for a disabled child for at least one year

Exclusion Criteria:

* Having more than one disabled child and being responsible for their care
* Having previously undergone surgery on the lower back
* Having a previous upper extremity disorder
* Receiving psychological treatment or medication
* Being pregnant or having recently given birth
* Having a recent history of trauma to the musculoskeletal system
* Having a defined chronic illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers of Children with Disabilities
Study Population: Mothers of Children with Disabilities
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
. Beck Depression Inventory | Baseline
  It is a scale consisting of 21 items that measures depressive symptoms. A maximum of 63 points can be obtained, with higher scores indicating an increase in depression.
Physical Workload Questionnaire | Baseline
  A 19-item Likert scale with scores ranging from 0 to 4, developed to identify the load on the lumbar region during work activities. Higher scores indicate increased work load.
Handgrip strength measurement | Baseline
  This measurement was performed on the dominant hand while the participant was seated in a chair in the standard position defined by the American Hand Therapy Association. They were asked to squeeze the dynamometer as hard as possible. The average of three measurements taken at 30-second intervals was recorded in pounds.

SECONDARY OUTCOMES:
1-10 Numerical Pain Rating Scale (NPRS) | Baseline
  The NPRS was used to determine the severity of low back pain reported at the time of assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No